CLINICAL TRIAL: NCT04299009
Title: Bright Light Therapy for Residual Daytime Symptoms Associated With Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: E3304-P; 1I21RX003304-01A1 (NIH)
Record Dates: First submitted 2020-03-02; First posted 2020-03-06 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: sleep apnea; CPAP; daytime sleepiness; bright light therapy
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Disorders of Excessive Somnolence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Retimer bright light therapy glasses (Experimental): active bright light therapy in the green/blue spectrum range
  Interventions: Device: Bright light therapy glasses
- sham-Retimer bright light therapy glasses (Sham Comparator): bright light therapy with light in the red spectrum (not active)
  Interventions: Device: Bright light therapy glasses

INTERVENTIONS:
Device: Bright light therapy glasses — Bright light therapy delivered through glasses
  Other Names: BLT

SUMMARY:
Sleep apnea is one of the most common chronic condition among US military Veterans, causing sleepiness, reduced psychomotor vigilance and depression, which undermine daytime functioning and quality of life. Persistent daytime symptoms of sleepiness in individuals with Obstructive Sleep Apnea (OSA) who are using Continuous Positive Airway Pressure (CPAP) are associated with adverse long term medical and functional outcomes. Residual daytime sleepiness (RDS) is associated with reduced occupational and family functioning and overall lower quality of life. Napping is a common behavior among individuals with OSA and RDS and has been linked to both benefits to and decline in health and functioning. Longer nap times may maintain, as opposed to decrease, sleepiness by promoting sleep inertia and can contribute to maintaining subclinical circadian alterations that result in higher night-tonight variability in sleep patterns. Preliminary studies in humans and animal models have shown persisting alterations of circadian rhythms in OSA patients, that fail to normalize with CPAP treatment. CPAP treatment, while effective at correcting respiratory events and night time blood oxygen saturation levels, does not necessarily re-align the circadian system. Current treatment options are limited to stimulants and modafinil, whose long-term safety profile, effectiveness and impact on functional recovery is largely unknown. Supplementary exposure to bright light has beneficial effects on sleep quality and daytime vigilance in healthy individuals and it has been increasingly applied in a variety of sleep and neuropsychiatric conditions. However, no study to date has tested the application of BLT to treat daytime symptoms associated with sleep apnea. The investigators' study will be the first to explore the role of Bright Light Therapy (BLT), a well-established non-pharmacological intervention for circadian disturbances, for the treatment of residual daytime symptoms of OSA which do not respond to CPAP.

DETAILED DESCRIPTION:
Due to COVID-19 pandemic emergency measures, recruitment for clinical trials is currently on hold

Background: Sleep apnea is one of the most common chronic condition among US military Veterans , it causes sleepiness, reduced psychomotor vigilance and depression, which undermine daytime functioning and quality of life . Persistent daytime symptoms of sleepiness and depression in individuals with OSA who are using Continuous Positive Airway Pressure (CPAP) are associated with adverse long term medical and functional outcomes . Current treatment options are limited to stimulants and modafinil, whose long-term safety profile, effectiveness and impact on functional recovery is largely unknown. The mechanisms for residual daytime symptoms in CPAP-treated sleep apnea are poorly understood and very little attention has been placed on interplay between sleep apnea and the circadian system. Notably, sleepiness, fatigue and depression, cardinal symptoms of OSA syndrome, are common manifestations of circadian misalignment. Circadian rhythms are synchronized to the environmental light or dark and to social activity cycles by zeitgebers (time givers) .Preliminary studies in humans and animal models have shown persisting alterations of circadian rhythms in OSA patients, that fail to normalize with CPAP treatment. CPAP treatment, while effective at correcting respiratory events and night time blood oxygen saturation levels, does not necessarily re-align the circadian system. Supplementary exposure to bright light has beneficial effects on sleep quality and daytime vigilance in healthy individuals and it has been increasingly applied in a variety of sleep and neuropsychiatric conditions. However, no study to date has tested the application of BLT to treat daytime symptoms associated with sleep apnea. The investigators' study will be the first to explore the role of Bright Light Therapy (BLT), a well-established non-pharmacological intervention for circadian disturbances, for the treatment of residual daytime symptoms of OSA which do not respond to CPAP.

ELIGIBILITY:
Inclusion Criteria:

* Veterans from the VA Pittsburgh Healthcare System (VAPHS)
* Documented diagnosis of OSA
* Currently on CPAP or BiPAP with documented adherence (defined as wearing CPAP/BiPAP for >4h/night on at least 75% of nights)
* Excessive residual daytime sleepiness (Epworth score > 10)
* Endorsing depressive symptoms (Quick Inventory of Depressive Symptomatology (Self-Report) [QIDS-SR] score>8)

Exclusion Criteria:

* Shift work
* Travel across time zones in the past month
* Narcolepsy
* Congestive heart failure (CHF)
* Poorly controlled diabetes (HgA1c>7%)
* Active substance use disorder
* Dementia
* Bipolar disorder

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabella Soreca, MD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soreca I, Arnold N, Dombrovski AY. Bright light therapy for CPAP-resistant OSA symptoms. J Clin Sleep Med. 2024 Feb 1;20(2):211-219. doi: 10.5664/jcsm.10840. PMID 37767823

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The available effective window for recruitment of participants was drastically reduced by the pandemic, during which all research activities and non essential clinical contact was place on hold
Groups:
- Sham-Bright Light Therapy (sBLT) First, Then BLT: Participants received sBLT therapy via Retimer glasses with a neutral density filter applied to the led lights, thus blocking 85% of the light intensity for 4 weeks, followed by BLT
- Bright Light Therapy (BLT) First, Then sBLT: Participants received BLT via Retimer glasses for 4 weeks, followed by 4 weeks of sBLT
Period: First Intervention (4 Weeks)
Arm/Group | Sham-Bright Light Therapy (sBLT) First, Then BLT | Bright Light Therapy (BLT) First, Then sBLT
Started | 9 | 6
Completed | 8 | 6
Not Completed | 1 | 0
Period: Second Intervention (4 Weeks)
Arm/Group | Sham-Bright Light Therapy (sBLT) First, Then BLT | Bright Light Therapy (BLT) First, Then sBLT
Started | 8 | 6
Completed | 8 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- sBLT Then BLT: sBLT first, followed by BLT
- BLT Then sBLT: BLT first, followed by sBLT
- Total: Total of all reporting groups
Arm/Group | sBLT Then BLT | BLT Then sBLT | Total
Number analyzed (Participants) | 9 | 6 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 6 | 15
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (5) | 54.8 (5) | 54.8 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 7 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 8 | 5 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Recruitment and Retention
Description: Number of participants recruited, number of participants retained, number of participants with complete data
Time Frame: baseline to week 9
Measure: Number; unit: participants
Groups:
- sBLT-BLT: sBLT first, followed by BLT
- BLT-sBLT: BLT first, followed by sBLT
Arm/Group | sBLT-BLT | BLT-sBLT
Number analyzed (Participants) | 9 | 6
participants
  Completers | 8 | 6
  Number of subjects with complete data | 8 | 6

2. Primary Outcome: Epworth Sleepiness Scale
Description: Brief self report questionnaire used to quantify degree of daytime sleepiness. Minimum score is 0,maximum score is 24; values below 10 are considered normal
Time Frame: pre- treatment=baseline; post-treatment=4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- sBLT: sham BLT for 4 weeks
- BLT, Active Treatment: BLT for 4 weeks,
Arm/Group | sBLT | BLT, Active Treatment
Number analyzed (Participants) | 14 | 14
score on a scale
  Epworth pretreatment | 13.2 (4) | 12.3 (4)
  Epworth post treatment | 12 (4.9) | 10.8 (4)
Statistical Analysis 1: Comparison: sBLT vs BLT, Active Treatment; Test type: Other — multilevel linear models with Epworth sleepiness score scores as the dependent variable; treatment block (BLT vs sBLT) as a fixed effect; treatment sequence as a covariate; and participant intercept as a random effect; p < 0.05, Mixed Models Analysis; regression coefficient = 2.45, 95% CI 2-sided [-0.30 to 5.19]

3. Secondary Outcome: Functional Outcomes of Sleep Questionnaire (FOSQ-10)
Description: Assesses impact of sleep related disturbances on daily functioning. It is a likert scale whose scaling of items is from zero to four. The potential range of scores for the total score is 5-20, with higher scores indicating worse functioning
Time Frame: pre-treatment=baseline; post-treatment=4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- BLT Active Treatment: BLT for 4 weeks,
Arm/Group | sBLT | BLT Active Treatment
Number analyzed (Participants) | 14 | 14
score on a scale
  FOSQ pre treatment | 24 (5) | 28.6 (3.2)
  FOSQ post treatment | 30 (5.3) | 29.5 (9)

ADVERSE EVENTS:
Time Frame: Each participants was assessed for a total of 10 weeks max from consent signing to end of the study.
Description: consistent with clinicaltrials.gov definition
Groups:
- Sham-Bright Light Therapy (sBLT): sham bright light therapy first, follow by one week wash out and them active bright light therapy
  Active treatment: Bright light therapy delivered through Retimer glasses. Sham treatment: neutral density filter blocking 80% of light intensity applied to Retimer glasses.
- Bright Light Therapy (BLT): active bright light therapy first, followed by one week wash out and then sham Bright light therapy Active treatment: Bright light therapy delivered through Retimer glasses. Sham treatment: neutral density filter blocking 85% of light intensity applied to Retimer glasses.
Arm/Group | Sham-Bright Light Therapy (sBLT) | Bright Light Therapy (BLT)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 1/14 | 1/14
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham-Bright Light Therapy (sBLT) (N=14) | Bright Light Therapy (BLT) (N=14)
Headache (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/09/NCT04299009/Prot_SAP_001.pdf
  • Informed Consent Form (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/09/NCT04299009/ICF_000.pdf